CLINICAL TRIAL: NCT03658304
Title: A Single Arm Phase II Trial of the Intraoperative Intravesical Instillation of Mitomycin C During Nephroureterectomy for Urothelial Carcinoma of the Upper Urinary Tract
Brief Title: Trial of Mitomycin C During Nephroureterectomy for Urothelial Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UF-GU-001; OCR18677 (Other: University of Florida); IRB201802090 (Other: University of Florida)
Record Dates: First submitted 2018-08-31; First posted 2018-09-05 (Actual); Results first posted 2022-11-02 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mitomycin C (Experimental)
  Interventions: Drug: Mitomycin c

INTERVENTIONS:
Drug: Mitomycin c — All participants will receive a single 40 mg dose of mitomycin C intraoperatively during their scheduled nephroureterectomy. This single dose will be given through a catheter in the subject's bladder.

SUMMARY:
Results of previous studies suggest that the timing of intravesical mitomycin C administration may impact bladder tumor recurrence rate following radical nephroureterectomy. This is the first study of its kind to attempt to identify the importance of timing of mitomycin C administration relative to bladder tumor recurrence rate following radical nephroureterectomy.This study will investigate the one year bladder tumor recurrence rate in patients with urothelial carcinoma of the upper urinary tract following intraoperative administration of mitomycin C during a nephroureterectomy, as well as the time to bladder tumor recurrence in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Both males and females ≥ eighteen years of age
* Clinical diagnosis of urothelial carcinoma of the renal pelvis and/or ureter. Clinical diagnosis of urothelial carcinoma may be based upon radiographic, pathologic or cytological findings alone or in combination with one another. No other histology is allowed.
* The TNM stage of the subject's disease (using the American Joint Committee on Cancer [AJCC] Cancer Staging Manual, 8th Edition) must be Tis, Ta, T1, T2, or T3, N0, M0. Subjects may have either a high-grade or low-grade tumor.
* ECOG performance status of 0-2
* Written informed consent obtained from the subject and the ability for the subject to comply with all the study-related procedures.
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy prior to and for at least 3 months after mitomycin C instillation to minimize the risk of pregnancy. Prior to study enrollment, women of childbearing potential must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy.
* Males with female partners of child-bearing potential must agree to use physician-approved contraceptive methods (e.g., abstinence, condoms, vasectomy) should avoid conceiving children prior to and for 3 months following mitomycin C instillation
* Subjects must have hemoglobin ≥ 9 g/dL and a platelet count ≥ 100,000/μL.

Exclusion Criteria:

* Active urothelial carcinoma of the bladder within 12 months prior to enrollment
* History of adverse reaction to mitomycin C
* Evidence of regional or metastatic disease.
* History of radical cystectomy
* Planned radical cystectomy at the time of nephroureterectomy
* Females or males of childbearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy prior to and for at least 3 months after mitomycin C instillation.
* Females who are pregnant or breastfeeding.
* History of any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of protocol therapy or that might affect the interpretation of the results of the study or that puts the subject at high risk for treatment complications, in the opinion of the treating physician.
* Prisoners or subjects who are involuntarily incarcerated.
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical illness.
* Subjects demonstrating an inability to comply with the study and/or follow-up procedures

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2023-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Crispen, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mitomycin C
Started | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Mitomycin C
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 25
Age, Continuous [Mean (Full Range); unit: years] | 70.14 [57 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 28
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Bladder Tumor Recurrence Rate
Description: The bladder tumor recurrence rate will be measured by the percentage of subjects who are confirmed by bladder biopsy to have a recurrence of urothelial carcinoma in the bladder following nephroureterectomy
Time Frame: 1 year
Population: all 29 subjects enrolled have reached the 1 year post-surgery timepoint.
Measure: Number; unit: percentage of subjects
Arm/Group | Mitomycin C
Number analyzed (Participants) | 29
percentage of subjects | 41.37

2. Secondary Outcome: Time to Bladder Tumor Recurrence
Description: Determine the median time to bladder tumor recurrence. A subject is considered to have had a bladder tumor recurrence when they have been confirmed by bladder biopsy to have a recurrence of urothelial carcinoma in the bladder following nephroureterectomy.
Time Frame: 3 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Mitomycin C
Number analyzed (Participants) | 29
days | 464 [210 to NA] — Upper confidence interval is not estimable because an insufficient number of subjects had a recurrence.

3. Secondary Outcome: Percentage of Subjects Who Had a Bladder Tumor Recurrence 3 Years Post-operatively
Description: Determine the percentage of subjects who are confirmed by bladder biopsy to have a recurrence of urothelial carcinoma in the bladder following nephroureterectomy 3 years post-operatively.
Time Frame: 3 years
Measure: Number; unit: percentage of subjects
Arm/Group | Mitomycin C
Number analyzed (Participants) | 29
percentage of subjects | 58.62

ADVERSE EVENTS:
Time Frame: Adverse event data were collected, at a minimum, from the time of informed consent until 30 days after mitomycin C instillation. Adverse event data were collected for a maximum of 1,057 days for all participants.
Description: Adverse events were assessed by the principal investigator, the treating sub-investigator, and/or the study coordinator from the time of informed consent until 30 days after mitomycin c instillation at a minimum. Adverse events were assessed by physical examination, labs, and subject self-reports.
Arm/Group | Mitomycin C
All-Cause Mortality (participants affected / at risk) | 4/29
Serious Adverse Events (participants affected / at risk) | 1/29
Other Adverse Events (participants affected / at risk) | 27/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mitomycin C (N=29)
Fever (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mitomycin C (N=29)
Vertigo (Ear and labyrinth disorders) | 1
Vomiting (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 4
Anemia (Blood and lymphatic system disorders) | 4
Wound complication (Injury, poisoning and procedural complications) | 1
Creatinine increased (Investigations) | 6
Edema limbs (General disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Dizziness (Nervous system disorders) | 2
Hematuria (Renal and urinary disorders) | 1
Hypercapnia (Blood and lymphatic system disorders) | 1
Hypotension (Vascular disorders) | 1
Melena (Gastrointestinal disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Delirium (Psychiatric disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Urinary tract infection (Infections and infestations) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Phlebitis (Blood and lymphatic system disorders) | 1
Urinary retention (Renal and urinary disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 2
Constipation (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Urine output decreased (Investigations) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Bloating (Gastrointestinal disorders) | 1
Cellulitis (Skin and subcutaneous tissue disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2
Pain (Surgical and medical procedures) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 1
White blood cell decreased (Investigations) | 1
Sinus tachycardia (Cardiac disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Chest pain (Cardiac disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
GI upset (Gastrointestinal disorders) | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Pruritis (Skin and subcutaneous tissue disorders) | 1
Urinary frequency (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-17): https://cdn.clinicaltrials.gov/large-docs/04/NCT03658304/Prot_SAP_000.pdf